CLINICAL TRIAL: NCT05125536
Title: The Effect of Music on Decreasing of Adaptation Difficulty in Alzheimer's Patients: Randomized Controlled Study
Brief Title: The Effect of Music in Alzheimer's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Munevver Kiyak, Instructor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AHMUGAE
Record Dates: First submitted 2021-10-22; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Music; Adaptation difficulty; Nursing care
MeSH Terms: conditions — Alzheimer Disease | interventions — Music Therapy; Rutin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Before the application, the "Descriptive Characteristics Data Form" and "Assessment Scale of Adaptation Difficulty in Elderly" were administered to the experimental group by the investigator through face-to-face interviews. A cd containing songs in Nihavent theme (instrumental), computer and sound system were used during the application. The patients in the experimental group were informed about the music session in advance. The sessions lasted 12 weeks in total and there were two sessions per week (Monday and Wednesday), and each session took approximately 50 minutes to complete. One week after the last music session (end of 12th week), the "Assessment Scale of Adaptation Difficulty in the Elderly" was re-administeredto the experimental group .
  Interventions: Other: Music therapy
- Control group (No Intervention): No intervention was performed for the patients in the control group.

INTERVENTIONS:
Other: Music therapy — rutin
  Other Names: rutin
  Arms: Experimental group

SUMMARY:
This study was randomized controlled study conducted to determine the effect of Nihavent theme on reducing adjustment difficulties in Alzheimer's patients.

The study was carried out with 30 patients.15 patients constituted the experimental group and 15 patients formed the control group. Before the application, the scale was administered to both groups through face-to-face interviews. The patients in the experimental group were informed about the music session in advance.Instrumental songs in nihavent theme were played with the sound system to the experimental group. The sessions were lasted 12 weeks in total and there were two sessions per week, and each session took approximately 50 minutes to complete. While no intervention was performed for the patients in the control group. One week after the last music session, the the scale was re-administered to both groups.

DETAILED DESCRIPTION:
Adaptation levels of Alzheimer's patients should be determined before planning nursing interventions. Institutions should support healthcare personnel in organizing music sessions for patients. It is believed that further studies examining the effect of the Nihavent theme in decreasing adaptation difficulty in Alzheimer's patients should be conducted with larger sample groups. The effects of verbal and non-verbal music on Alzheimer's patients should also be evaluated and compared to gain further insight on this important matter.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 age range
* Were conscious able to communicate and active

Exclusion Criteria:

* Change in their diagnosis, medications, consciousness, and/or drug dose
* During the study period they a regression in emotional state (crying, sadness)
* Those with complex diseases such as cancer

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Assessment Scale of Adaptation Difficulty for Elderly | 24 days
  This scale was developed by Şişman et al. in 2016 in order to determine the adaptation of elderly individuals, and its validity and reliability were determined. Chronbach alpha internal consistency coefficient was found to be 0.93. It is a likert-type scale consisting of 24 questions. The answers to each item were determined as 0 points for "never", 1 point for "some", 2 points for "quite a lot" and 3 points for "a lot". The scores obtained from the items in the scoring of the scale are calculated by summing and dividing by the number of questions. The average score that can be obtained from the scale is 0 points as the lowest and 3 points at the highest. As the individual's score from the scale decreases, the level of compliance increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No